CLINICAL TRIAL: NCT04365049
Title: Nab-Paclitaxel and Gemcitabine Plus Camrelizumab and Radiotherapy Versus Nab-Paclitaxel and Gemcitabine Alone for Locally Advanced Pancreatic Adenocarcinoma
Brief Title: Nab-Paclitaxel and Gemcitabine Plus Camrelizumab and Radiotherapy for Locally Advanced Pancreatic Adenocarcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Ming Kuang, The vice president, Sun Yat-sen University
Other Study IDs: HepBilPan001
Record Dates: First submitted 2020-04-24; First posted 2020-04-28 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: PDAC - Pancreatic Ductal Adenocarcinoma
MeSH Terms: interventions — Radiotherapy; 130-nm albumin-bound paclitaxel; Gemcitabine; camrelizumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nab-Paclitaxel+Gemcitabine+Camrelizumab+Radiotherapy: Chemotherapy consisted of eight 21-day cycles of nab-paclitaxel plus gemcitabine (nab-paclitaxel 125 mg/m² by intravenous infusion for approximately 30-45 mins, followed by gemcitabine 1000mg/m² intravenous infusion for approximately 30 mins on days 1 and 8). Anti-PD-1 antibody (camrelizumab, Hengrui Medicine Co., Ltd) 200 mg was administered intravenously for 30 mins every three weeks. During the chemotherapy-treated period, camrelizumab was administered on day 1 of each 21-day cycle before the infusion of chemotherapy. Radiotherapy started after two cycles of chemotherapy. A total radiation dose greater than 50 Gy without damaging organ function was the essential requirement.
  Interventions: Radiation: Radiotherapy; Drug: Nab-paclitaxel; Drug: Gemcitabine; Drug: Camrelizumab
- Nab-Paclitaxel+Gemcitabine: Chemotherapy consisted of eight 21-day cycles of nab-paclitaxel plus gemcitabine (nab-paclitaxel 125 mg/m² by intravenous infusion for approximately 30-45 mins, followed by gemcitabine 1000mg/m² intravenous infusion for approximately 30 mins on days 1 and 8).
  Interventions: Drug: Nab-paclitaxel; Drug: Gemcitabine

INTERVENTIONS:
Radiation: Radiotherapy — Radiotherapy started after two cycles of chemotherapy. External beam radiation therapy was performed using an intensity modulated radiation therapy technique. The gross target volume included the gross primary tumor and positive regional lymph nodes as defined by the multiphasic imaging. A total radiation dose greater than 50 Gy without damaging organ function was the essential requirement.
  Groups: Nab-Paclitaxel+Gemcitabine+Camrelizumab+Radiotherapy
Drug: Nab-paclitaxel — Eight 21-day cycles of nab-paclitaxel 125 mg/m² by intravenous infusion for approximately 30-45 mins on days 1 and 8.
Drug: Gemcitabine — Eight 21-day cycles of gemcitabine 1000mg/m² intravenous infusion for approximately 30 mins on days 1 and 8.
Drug: Camrelizumab — Anti-PD-1 antibody (camrelizumab, Hengrui Medicine Co., Ltd) 200 mg was administered intravenously for 30 mins every three weeks. During the chemotherapy-treated period, camrelizumab was administered on day 1 of each 21-day cycle before the infusion of chemotherapy.
  Groups: Nab-Paclitaxel+Gemcitabine+Camrelizumab+Radiotherapy

SUMMARY:
The study is a prospective and observational cohort study. The purpose is to to investigate the safety and efficacy of nab-paclitaxel and gemcitabine plus camrelizumab and radiotherapy versus nab-paclitaxel and gemcitabine alone for locally advanced pancreatic adenocarcinoma (PDAC)

DETAILED DESCRIPTION:
We will prospectively collect 100 patients who receive nab-paclitaxel and gemcitabine plus camrelizumab and radiotherapy or nab-paclitaxel and gemcitabine alone. Data will be stored in a private database. The process of data collection will be supervised and regular data examination will be performed.

ELIGIBILITY:
Inclusion Criteria:

1. aged 18-75 years;
2. histologically or cytologically proven diagnosis of pancreatic adenocarcinoma;
3. treatment-naive locally advanced pancreatic cancer (locally advanced status was determined by our multidisciplinary team based on the National Comprehensive Cancer Network definitions);
4. no distant metastasis as defined by CT or MRI of the chest, abdomen and pelvis;
5. at least 1 measurable lesion based on the Response Evaluation Criteria in Solid Tumors criteria (RECIST) 1.1;
6. an Eastern Cooperative Oncology Group (ECOG) performance status score of 0 to 1;
7. adequate hematological, liver, renal function:

   1. absolute neutrophil count≥1500 cell/mm3;
   2. platelet count≥100×109/L;
   3. hemoglobin concentration >90 g/L;
   4. albumin≥30 g/L ;
   5. total bilirubin<1.5 times the upper limit of normal;
   6. alanine aminotransferase and aspartate aminotransferase≤3 times the upper limit of normal;
   7. serum creatinine concentration<1.5 times the upper limit of the normal range or less and creatinine clearance rate≥45 mL/min;
8. life expectancy of at least 3 months.

Exclusion Criteria:

1. with any other malignancy within the 5 years before enrolment;
2. with active infections (bacterial, viral, or fungal) requiring systematic treatment, with hepatitis B or C infection, or a history of HIV infection, or receiving immunosuppressive therapy;
3. with peripheral sensory neuropathy at a grade >1;
4. with a history of allergy or hypersensitivity to the study drugs;
5. pregnant or breast feeding women, reproductive aged women who refused to take adequate contraceptive measures during the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Advanced Pancreatic Adenocarcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-04-01 (Actual); Primary Completion 2023-12 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | two years
  defined as the time from randomization until disease progression or death from any cause, whichever happens first. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive and progression free. Patients not having an event will be censored at the date last seen alive.
Overall survival | two years
  defined as the time from randomization until death from any cause. Patients who withdraw or who are lost to follow-up will be censored at the date last known to be alive. Patients remaining alive throughout the duration of the study will have their survival time censored on the date last seen alive.

SECONDARY OUTCOMES:
Adverse events | two years
  adverse events during the treatment period using Common Terminology Criteria for Adverse Events (CTCAE) (version 5.0).
Tumor response | two years
  measured according to the Response Evaluation Criteria in Solid Tumors (RECIST) criteria 1.1 by means of computed tomography (CT) or magnetic resonance imaging (MRI) at each follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ming Kuang, PhD, Study Chair — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- Frist Affliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China